CLINICAL TRIAL: NCT06634875
Title: A Phase IIa, Non-Randomized, Open-Label Dose Expansion Trial of Isunakinra in Combination With Pembrolizumab in Patients With Metastatic or Unresectable, Locally Advanced Colorectal Cancer
Brief Title: Isunakinra Alone and in Combination With Pembrolizumab in Patients With Colorectal Cancer (MSS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Buzzard Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUZ02CD101
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colorectal cancer; microsatellite stable; MSS; kras mutated; TMB-H; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — EBI-005

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- combination immunotherapy (Experimental)
  Interventions: Drug: isunakinra

INTERVENTIONS:
Drug: isunakinra — Isunakinra is a potent IL1R1 inhibitor
  Other Names: EBI-005

SUMMARY:
This study will enroll patients with colorectal cancer that is locally advanced or metastatic. The tumor must be microsatellite stable (MSS), have a tumor mutational burden that is high (TMB-H) and be kras mutated. Patients must have been treated with available approved treatments already. In this study the investigators are testing a new type of immunotherapy, the potent IL-1 inhibitor isunakinra to be added to already approved immunotherapy (PD-1/PD-L1 inhibitor) in an attempt to get this treatment to work in this treatment resistant type of tumor.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must have:

  * Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum

    * Tumor is determined to be RAS-mutated (KRAS, NRAS or HRAS) and microsatellite stable/proficient in mismatch repair, as assessed by immunohistochemistry (IHC) and/or polymerase chain reaction (PCR)/next generation sequencing (NGS) in a Clinical Laboratory Improvement Act (CLIA) environment and with a tumor mutational burden (TMB) of 10 MB or more.

      2. The study patients are required to have measurable disease by radiographic criteria (RECIST 1.1 and iRECIST).

      3. Prior therapy: Patients must have completed or had disease progression on at least one prior line of disease-appropriate therapy for metastatic disease (with or without PD-1 inhibitors), with no available therapy likely to convey clinical benefit, or not be candidates for therapy of proven efficacy for their disease.

      4. There should be a minimum of 4 weeks from any prior chemotherapy (except for the nitrosoureas and mitomycin C, requiring a minimum of 6 weeks), immunotherapy and/or radiation. Patients with prostate cancer on hormone deprivation therapy may continue that therapy while on study.

      5. Patients must have recovered (grade 1 or baseline) from any clinically significant toxicity associated with prior therapy (for example, alopecia is not clinically significant).

      6. ECOG performance status ≤ 1 7. Patients must have normal organ and hematologic function as defined below:
    * Serum creatinine ≤ 1.5 x upper limit of normal OR creatinine clearance and a 24-h urine collection of ≥ 60 mL/min.
    * ALT and AST ≤ 3x the upper limits of normal.
    * Total bilirubin ≤ 1.5 x upper limit of normal OR in patients with Gilbert's syndrome, a total bilirubin ≤ 3.0.
    * Hematological eligibility parameters (within 16 days of starting therapy):

      * Granulocyte count ≥ 1,500/mm3
      * Platelet count ≥ 75.000/mm3 8. Patients must have baseline pulse oximetry > 90% on room air at rest.

Exclusion Criteria:

1. Subjects must have:

   ⦁ Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum

   • Tumor is determined to be RAS-mutated (KRAS, NRAS or HRAS) and microsatellite stable/proficient in mismatch repair, as assessed by immunohistochemistry (IHC) and/or polymerase chain reaction (PCR)/next generation sequencing (NGS) in a Clinical Laboratory Improvement Act (CLIA) environment and with a tumor mutational burden (TMB) of 10 MB or more.
2. The study patients are required to have measurable disease by radiographic criteria (RECIST 1.1 and iRECIST).
3. Prior therapy: Patients must have completed or had disease progression on at least one prior line of disease-appropriate therapy for metastatic disease (with or without PD-1 inhibitors), with no available therapy likely to convey clinical benefit, or not be candidates for therapy of proven efficacy for their disease.
4. There should be a minimum of 2 weeks wash out period from chemotherapy and/or radiation therapy, and 4 weeks wash out period for immunotherapy.
5. Patients must have recovered (grade 1 or baseline) from any clinically significant toxicity associated with prior therapy (for example, alopecia is not clinically significant).
6. ECOG performance status ≤ 1
7. Patients must have normal organ and hematologic function as defined below:

   * Serum creatinine ≤ 1.5 x upper limit of normal OR creatinine clearance and a 24-h urine collection of ≥ 60 mL/min.
   * ALT and AST ≤ 3x the upper limits of normal.
   * Total bilirubin ≤ 1.5 x upper limit of normal OR in patients with Gilbert's syndrome, a total bilirubin ≤ 3.0.
   * Hematological eligibility parameters (within 16 days of starting therapy):

     * Granulocyte count ≥ 1,500/mm3
     * Platelet count ≥ 75.000/mm3
8. Patients must have baseline pulse oximetry > 90% on room air at rest.

Exclusion criteria

1. Pregnant women or women presently breast-feeding their children are excluded due to unknown risks to a developing fetus or infant, confirmed by negative pre-treatment serum pregnancy test.
2. Concurrent treatment for cancer, with specific exceptions noted in inclusion criteria.
3. Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
4. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
5. Active autoimmune diseases requiring treatment. However, patients with vitiligo, alopecia, or clinically stable autoimmune endocrine disease who are on stable dosing of appropriate replacement therapy (if such therapy is indicated) are eligible.
6. Concurrent use of systemic steroids, except for physiologic doses of systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited pharmacologic doses of systemic steroids (e.g., in patients with exacerbations of reactive airway disease or to prevent iv contrast allergic reaction or anaphylaxis in patients who have known contrast allergies) are allowed.
7. Patients who are receiving any other investigational agents within 28 days before start of study treatment.
8. Patients with untreated central nervous system metastases or local treatment of brain metastases within the last 2 months. Patients with stable brain metastasis for 2 months post-intervention are eligible.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or any of its excipients or a history of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in study.
10. Serious or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
11. HIV-positive patients are ineligible because of the potential for decreased immune response.
12. Patients unwilling to use adequate contraception (defined as hormonal or barrier method or abstinence) prior to study entry are excluded. If the patient needs to be on adequate contraception, contraception must start before study entry and continue for 3 months after completion of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 months
  The incidence, relatedness and severity of adverse events (includes safety laboratory abnormalities) per CTCAE v. 5
PFS | 6 months
  Progression Free Survival per iRECIST

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - USC/Norris Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kovalchin J, King B, Masci A, Hopkins E, Fry J, Hou J, Li C, Tenneson K, Weber S, Wolfe G, Collins K, Furfine ES. Preclinical Development of EBI-005: An IL-1 Receptor-1 Inhibitor for the Topical Ocular Treatment of Ocular Surface Inflammatory Diseases. Eye Contact Lens. 2018 May;44(3):170-181. doi: 10.1097/ICL.0000000000000414. PMID 28727604
- [Background] Hou J, Townson SA, Kovalchin JT, Masci A, Kiner O, Shu Y, King BM, Schirmer E, Golden K, Thomas C, Garcia KC, Zarbis-Papastoitsis G, Furfine ES, Barnes TM. Design of a superior cytokine antagonist for topical ophthalmic use. Proc Natl Acad Sci U S A. 2013 Mar 5;110(10):3913-8. doi: 10.1073/pnas.1217996110. Epub 2013 Feb 19. PMID 23431173
- [Background] Spella M, Ntaliarda G, Skiadas G, Lamort AS, Vreka M, Marazioti A, Lilis I, Bouloukou E, Giotopoulou GA, Pepe MAA, Weiss SAI, Petrera A, Hauck SM, Koch I, Lindner M, Hatz RA, Behr J, Arendt KAM, Giopanou I, Brunn D, Savai R, Jenne DE, de Chateau M, Yull FE, Blackwell TS, Stathopoulos GT. Non-Oncogene Addiction of KRAS-Mutant Cancers to IL-1beta via Versican and Mononuclear IKKbeta. Cancers (Basel). 2023 Mar 20;15(6):1866. doi: 10.3390/cancers15061866. PMID 36980752